CLINICAL TRIAL: NCT06023888
Title: A Prospective Randomized Controlled Study on the Waveform Periodicity Analysis of Complex Fractionated Electrograms With OctaRay in Patients With Persistent Atrial Fibrillation
Brief Title: Waveform Periodicity Analysis in Patients With Persistent Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chin-Yu Lin, Doctor, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-12-009C
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: persistent atrial fibrillation; ablation; driver
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This study was designed to determine the efficacy of substrate ablation using waveform periodicity analysis, similarity analysis with OCTARAY™ Mapping Catheter could collected more AF electrogram and facilitate the mapping resolution and driver identification., plus phase mapping in persistent AF patients who required substrate modification.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodicity-based (Experimental)
  Interventions: Other: Mapping strategy
- Control (Other): Standard ablation strategy as usual
  Interventions: Other: Mapping strategy

INTERVENTIONS:
Other: Mapping strategy — The ablation strategy was based on the mapping results of periodicity.
  Arms: Periodicity-based
Other: Mapping strategy — PVI+ non-PV trigger
  Arms: Control

SUMMARY:
STUDY DESIGN A prospective study.

OBJECTIVE A single center clinical trial on the analysis of intracardiac atrial electrogram waveform periodicity for catheter ablation of persistent atrial fibrillation with OCTARAY™ Mapping Catheter, as prospective randomized controlled study.

HYPOTHESIS:

The critical atrial substrates in maintaining persistent atrial fibrillation could be identified by non-linear electrogram morphology analysis in a point-by-point electroanatomic mapping. Based on the previous study, atrial substrate with high-similarity electrogram regions correlated with procedural AF termination and better long-term AF-free (1). Therefore, we proposed that the degree of waveform similarity plus the beat-to-beat sequential morphology (2) (duration of how many similar waveforms can maintain in sequence) would be even better to characterize the atrial substrate and could be potentially critical atrial substrate in prediction of sources of AF. As additional substrate mapping provided benefits compared to PVI alone in patients with persistent AF, we hypothesize that waveform periodicity adjuvant to electrogram similarity and phase mapping could be used to guide radiofrequency ablation in real time. The used of the OCTARAY™ Mapping Catheter could collected more AF electrogram and facilitate the mapping resolution and driver identification.

ELIGIBILITY:
Inclusion Criteria:

* persistent atrial fibrillation
* refractory or intolerant to medication

Exclusion Criteria:

* Previous AF ablation
* LA thrombus
* Previous MAZE procedure
* Poor renal function
* Can't follow-up for one year

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia | up to 6 month
  atrial arrhythmia in 24-hour monitoring
Recurrence of atrial arrhythmia | up to 1 year
  atrial arrhythmia in 7-day ECG monitoring(RootiRx®)
  The RootiRx® multi-sensor patch-type system is a water-resistant compact ECG patch of 62 × 22 × 9mm size and 14g of weight. It is applied on the patient left chest similar to lead II location and it is fixed on a disposable self-adhesive patch then connected to the skin with two electrodes. RootiRx Syste can make continuous ECG monitoring up to seven days at a sampling frequency of 250Hz with 24-bit high resolution. Proprietary algorithms are used to analyze recorded data.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan